CLINICAL TRIAL: NCT04373824
Title: To Study the Effectiveness of Ivermectin With Standard of Care Treatment Versus Standard of Care Treatment for COVID 19 Cases. A Pilot Study
Brief Title: Max Ivermectin- COVID 19 Study Versus Standard of Care Treatment for COVID 19 Cases. A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Max Healthcare Insititute Limited (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MHC-COVID-19- INV- ACT-BHR
Record Dates: First submitted 2020-04-26; First posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-05

CONDITIONS: COVID
MeSH Terms: interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: 25 subjects in each Arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I- Ivermectin (Experimental): First group with 25 confirmed cases of COVID 19 shall be treated with Ivermectin 200 to 400mcg per kg body weight on day 1 and day 2 along with standard treatment of the hospital protocol
  Interventions: Drug: Ivermectin
- Group II- standard treatment (No Intervention): The second group with 25 confirmed cases of COVID 19 shall be treated with standard treatment as per hospital protocol for COVID 19.

INTERVENTIONS:
Drug: Ivermectin — Ivermectin 200 to 400 mcg per kg body weight
  Arms: Group I- Ivermectin

SUMMARY:
At present, there are no specific treatments for COVID-19. WHO recommends four treatments for COVID 19 with drugs i.eRemdesivir, Lopinavir/ ritonavir, Lopinavir/ ritonavir with interferon beta -1a, and chloroquine or hydroxychloroquine. Currently, there are several ongoing clinical trials evaluating potential treatments. Recently, LeonCaly reported that Ivermectin, an FDA-approved anti-parasitic previously shown to have broad-spectrum anti-viral activity in vitro, is an inhibitor of the causative virus (SARS-CoV-2), with a single addition to Vero-hSLAM cells 2 hours post infection with SARSCoV-2 able to effect about 5000-fold reduction in viral RNA at 48 h. Ivermectin therefore warrant further investigation for possible benefits in humans. The study rationale is to understand the effect of the drug on eradication of virus.

DETAILED DESCRIPTION:
This study aims to confirm the antivirus effectiveness of Ivermectin on coronavirus i.e COVID 19 then to explore its potential use in the combating to the COVID 19 pandemics.

Enrollment of subject into the trial shall only occur after providing written permission to voluntarily participate into the study by signing and dating the informed consent form before starting any trial related treatment. 50 cases of COVID-19 will be enrolled into the trial. The trial shall be divided into two groups. First group with 25 confirmed cases of COVID 19 shall be treated with Ivermectin 200 to 400 mcg per kg body weight on day 1 and day 2 along with standard treatment of the hospital protocol. The second group with 25 confirmed cases of COVID 19 shall be treated with standard treatment as per hospital protocol for COVID 19. Subjects in both the arms shall be followed up for recovery of death with regular monitoring as per below schedule.

1. Test for virus at 1, 3 & 5 days from beginning of trial drug started for the patient in the hospital
2. Clinical profile of the patient every day of hospitalization
3. Investigation of pulmonary function and oxygen saturation every day of hospitalization
4. The day a patient is put on ventilator and the day when removed
5. The day a patient develops acute respiratory distress syndrome and the day when relieved All the above data shall be collected on paper case record form for interim and final analysis from start of the trial i.e enrollment, treatment and follow-up. Viral test to monitor the eradication of Virus shall be done free of cost from third day of enrollment and providing the study drug on daily basis upto eradication of virus or completion of the trial

ELIGIBILITY:
Inclusion Criteria:

1. Subjects within age group between 18 to 75 years
2. With either sex, male or female
3. Confirmed case of COVID-19 at Max Hospitals.

Exclusion Criteria:

* Patients who are critically sick

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04-25 (Actual); Primary Completion 2020-07-25 (Estimated); Study Completion 2020-07-25 (Estimated)

PRIMARY OUTCOMES:
effect of Ivermectin on eradication of virus. | 3 months
  Test for virus at 1, 3 & 5 days from beginning of trial drug started for the patient in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Budhiraja, MRCP, FACP, Principal Investigator — Max Healthcare
Locations (1):
- Max Super Speciality hospital, Saket (A unit of Devki Devi Foundation), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No